CLINICAL TRIAL: NCT00908063
Title: A Randomized, Placebo Controlled, Double-Blind, Single Dose, Dose Escalation Study to Evaluate the Safety and Tolerability of Oxycyte in Patients With Severe Non-Penetrating Traumatic Brain Injury
Brief Title: Safety and Tolerability of Oxycyte in Patients With Traumatic Brain Injury (TBI)
Acronym: STOP-TBI
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: futility
Sponsor: Tenax Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OX-CL-II-005
Record Dates: First submitted 2009-05-22; First posted 2009-05-25 (Estimated); Last update posted 2014-11-13 (Estimated); Status verified 2014-03

CONDITIONS: Traumatic Brain Injury
Keywords: TBI; Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — perfluoro(t-butylcyclohexane); Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oxycyte (Experimental): Single intravenous infusion of Oxycyte (Perfluoro(t-butylcyclohexane) Intravenous Emulsion 60% w/v)
  One of three volume doses based on cohort assignment (1.0 mL/min; 2.0 mL/min; 3.0 mL/min). The infusion will be administered at a rate of 15mL/min and will begin within 12 hours of injury.
  Interventions: Drug: Oxycyte
- Normal Saline (Placebo Comparator): Single intravenous infusion of Normal Saline
  One of three volume doses based on cohort assignment (1.0 mL/min; 2.0 mL/min; 3.0 mL/min). The infusion will be administered at a rate of 15mL/min and will begin within 12 hours of injury.
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Oxycyte — A single dose of one of three dosage levels (dose escalating design), given by intravenous infusion at the rate of 15 mL/min (total duration expected to be between 5 and 20 minutes).
  Other Names: Oxycyte Perfluoro(t-butylcyclohexane) Intravenous Emulsion 60% w/v
  Arms: Oxycyte
Drug: Normal Saline — Normal saline will be administered as one of three volume doses based on cohort assignment (1.0 mL/min; 2.0 mL/min; 3.0 mL/min). The infusion will be administered at a rate of 15mL/min and will begin within 12 hours of injury.
  Other Names: Placebo
  Arms: Normal Saline

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of a single administration of Oxycyte in patients with severe non-penetrating traumatic brain injury (TBI).

In the first dose level (Cohort 1), 11 patients were randomized 2:1 to receive either 1.0 mL/kg Oxycyte (0.6 g/kg; n=8) or NS (n=3). A total of 8 patients received Oxycyte. The Data Safety Monitoring Board (DSMB) reviewed the safety data for patients in Cohort 1 through Day 14, and approved escalation to the next dose.

In Cohort 2, 18 patients will be randomized 2:1 to receive either 2.0 mL/kg Oxycyte (1.2 g/kg; n=12) or NS (n=6). The DSMB will then review the safety data for all patients in Cohort 2 through Day 14 and either approve escalation to the highest dose or remain at the current dose. If remaining at the current dose level (Cohort 2) an additional 50 patients will be randomized 1:1 to Oxycyte (n=25) or NS (n=25) and treated.

If escalation occurs to Cohort 3, 18 patients would be randomized 2:1 to Oxycyte (n=12) or NS (n=6) to receive the 3.0 mL/kg dose. The DSMB would again review the safety data and decide whether to treat an additional 50 patients at this dose or to decrease the dose back to 2.0 mL/kg. This group would be randomized 1:1 to receive Oxycyte (n=25) or NS.

DETAILED DESCRIPTION:
This is a randomized, placebo controlled, double-blind, single dose, dose-escalation study to evaluate the safety and tolerability of Oxycyte in patients with severe non-penetrating Traumatic Brain Injury administered in conjunction with 50% to 80% oxygen and standard of care treatment.

At each dose level, patients receiving Oxycyte will be compared to a control group of patients who will receive Normal Saline (NS); all patients will receive 50% oxygen or greater, if per standard of care for a particular patient based on his / her condition, up to a maximum of 80%.

Ischemic brain damage is found in 80% of patients who die from severe head injury and studies have shown that early, transient cerebral hypoperfusion of unknown origin is present in about 40% of these patients. In several early research studies, it is documented that about one-third of severe head injured patients have reduced brain oxygen tension (<25 mm Hg) especially during the first 6 to 12 hours following severe head injury. In this group of patients with low brain oxygen, the clinical prognosis is poor with death being a frequent outcome.

Based on a belief that increased brain oxygen levels would prove beneficial in the TBI patient, it is theorized that perfluorocarbon-enhanced oxygen delivery may provide the same or greater benefit. PFCs are especially attractive in this setting for several reasons; first, because they transport oxygen without the need for erythrocytes and hemoglobin and can thus perfuse and oxygenate "peri-contusional" brain tissue in which it has been shown that capillaries are so narrowed as to impede red blood cell (RBC) transport; secondly, perfluorocarbon (PFCs) actually increase oxygen transport and oxygen tension in the tissues, which cannot be achieved with normobaric hyperoxia alone.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 - 70 years of age (inclusive) at the time of study entry
* Weight ≥45 kg
* Able to begin the infusion of study drug within 12 hours of injury
* Evidence of severe non-penetrating traumatic brain injury by clinical evaluation, clinical indication for intracranial pressure (ICP) monitoring, Glasgow Coma Scale (GCS) assessment (4-8 prior to randomization, obtained any time prior to dosing and including patients who deteriorate to severe TBI after arrival in the hospital, not including times when the patient is pharmacologically paralyzed for management or treatment) and with definite anatomic signs of injury on head CT scan (e.g., Marshall Grade II-VI or equivalent)
* At least one reactive pupil at screening. Just prior to study drug administration pupil reactivity must be confirmed again. If the patient is in the peri-postoperative period at that time and reactivity is difficult to assess due to small pupil size, the Investigator will determine if the patient is eligible based on clinical presentation.
* If a patient, due to his or her injuries is unable to provide written informed consent, then written consent may be obtained by an appropriate surrogate decision maker in accordance with preapproved procedures in compliance with local regulations.

Exclusion Criteria:

Patients who meet any of the following criteria will not be included in the study:

Physical Assessment:

* Not expected to survive the next 24 hours
* Morbidly obese (BMI >40)
* Absence of a motor response (not including times when the patient is pharmacologically paralyzed for management or treatment)
* Severe unexpected hyperthermia on admission (e.g. >39°C)
* Bilaterally fixed and dilated pupils
* Penetrating traumatic brain injury
* Major liver, kidney, or cardiac injury requiring operative intervention
* Major pulmonary injury, including lung contusion, severe atelectasis, acute respiratory distress syndrome, or acute aspiration pneumonitis
* Severe chronic obstructive pulmonary disease (COPD), pulmonary edema, or congestive heart failure in the judgment of the Investigator

Laboratory Values:

* Platelet count <100,000/mm3 at screening, prior to transfusion of any platelets
* Neutrophil count <1500 /mm3 at screening
* In the judgment of the Investigator, any clinically significant prolonged clotting time on INR, prothrombin time (PT) or activated partial thromboplastin time (aPTT), or any other coagulation test performed
* One or more of the following liver function test results: Total Bilirubin >2 x upper limit of normal (ULN), ALT >2.5 x ULN, or AST 2.5 > x ULN
* Women with a positive pregnancy test or known to be currently breastfeeding at screening

Concomitant Medications:

* Known use of immunosuppressive therapy (e.g. TNF inhibitors, methotrexate, cyclosporine, etc.)
* Concurrent use of Plavix® (clopidogrel bisulfate), Pradaxa® (dabigatran elexilate) or an anti- coagulant other than ≤100 mg/day aspirin for any condition

Known Medical History:

* Immersion injury
* Cardiopulmonary resuscitation (chest compression and/or external cardiac shock) required following the current injury
* Hemodynamically unstable (e.g., requiring >6L colloid or crystalloid fluid as well as >4 units of packed cells within 4 hours prior to enrollment)
* Known or suspected brain tumor
* Known severe allergy to any component of Oxycyte or known severe allergy to eggs
* Known to be immunocompromised (e.g. known history of HIV)
* Known history of major liver disease (e.g., liver failure, necrosis or cirrhosis) or chronic hepatitis B virus (HBV) or hepatitis C virus (HCV) infection
* Any known hematological or coagulopathic disorder that, in the Investigator's opinion, is likely to significantly impair platelet function or coagulation (e.g., hemophilia, von Willebrand's disease, myelodysplastic syndrome)
* History of severe TBI (previous to the current TBI) or any prior cerebral injury that required hospitalization and that may, in the Investigator's opinion, interfere with the results of this study
* Known history of any of the following diseases: Parkinson's disease, Huntington's disease, major stroke, seizure disorder, multiple sclerosis or cerebral aneurysm (unless clipped and stable, in which case patient may be included)
* Any life threatening condition prior to the current injury or other diseases or disorders that, in the Investigator's opinion, may put the patient at undue risk or confound the results of the study (e.g signs of soft tissue or other active infection)
* Current participation in another clinical trial with an investigational product, or participation in such a clinical trial within 30 days prior to screening
* Patients serving in the military forces at the time of screening who (if required) do not have the necessary approval from the appropriate authorities

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2009-10; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability will be compared between treatment groups as measured by frequency, severity, and type of adverse events and serious adverse events between treatment groups. | Through Day 30 or hospital discharge

SECONDARY OUTCOMES:
Efficacy as determined by short-term improvement | Through Day 7, 30, Month 3, and Month 6
  Short-term improvement will be compared between treatment groups as assessed by:
  * Functional outcomes as measured by the Glasgow Outcome Scale-Extended (GOSE)
  * Time to extubation
  * Time to intensive care unit (ICU) discharge and
  * Time to hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Michael Reinert, MD, Principal Investigator — Neurosurgery, Ospedale Regionale Lugano
Locations (6):
- Israel (5):
  - Soroka Medical Center, Beersheba, Ben Gurion
  - Rambam Health Care Campus, Haifa
  - Hadassah Medical Center, Jerusalem
  - Sheba Medical Center, Ramat Gan
  - Tel-Aviv Sourasky Medical Center, Tel Aviv
- Ospedale Regionale Lugano, Lugano, Switzerland